CLINICAL TRIAL: NCT05046782
Title: Abbreviated Biparametric MRI (RSI + T2WI) for Prostate Cancer Detection: Correlation With Histopathology
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn prior to full implementation due to logistical and resource-related considerations. Study procedures are currently under review and a new protocol may be considered pending the outcome of this review
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0823; NCI-2021-09145 (Other: NCI CTRP-Clinical Trials Gov Registry)
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI technique (Experimental): restriction spectrum imaging (RSI) can detect prostate cancer better than a standard-of-care MRI.
  Interventions: Device: restriction spectrum imaging (RSI)

INTERVENTIONS:
Device: restriction spectrum imaging (RSI) — detect prostate cancer better than a standard-of-care MRI

SUMMARY:
Multiparametric MRI of the prostate (mpMRI) plays an integral role in contemporary prostate cancer management. It involves the acquisition of both anatomical sequences (T1- and T2-weighted images) as well as 'functional' imaging sequences (diffusion weighted imaging (DWI) and dynamic contrast enhanced (DCE) imaging), the latter sequences being those which image water diffusivity and tissue perfusion, respectively. Advantages of mpMRI include ability to risk stratify patients prior to biopsy, enhanced detection of clinically significant cancer and reduced diagnosis of insignificant cancers, the identification of active surveillance candidates and improved local staging for subsequent surgical and radiotherapy planning. However, there are ongoing challenges encountered with prostate mpMRI in terms of patient acceptance, image acquisition technical challenges, interpretive expertise and cost.

These challenges have motivated recent investigations employing tailored MRI protocols, i.e. faster and less expensive MR exams that eliminate one or more aspects of current mpMRI technique considered redundant, while retaining the essential imaging parameters needed for equivalent diagnostic interpretation. Among these is non-contrast biparametric MRI, which involves anatomic T2 weighted images along with diffusion weighted images (DWI) as the only retained functional sequence. Both single center studies and meta analyses have demonstrated no added value for DCE compared to the combination of T2WI and DWI, Overall cancer detection rates have been found to be equivalent for bpMRI compared to mpMRI, independent of reader experience, with comparable efficacy to guide cognitive targeted, MRI-targeted and MRI-US fusion guided biopsy. Equivalence between bpMRI and mpMRI for cancer detection has also been corroborated in two recently published meta analyses. Based upon our institution's experience with prostate mpMRI, avoidance of gadolinium and DCE imaging would be associated with a 30 percent reduction in scan cost and 40 percent reduction in total time (i.e. scan time plus patient preparatory time).

DETAILED DESCRIPTION:
Primary Objective

This is a prospective study of men presenting to MD Anderson with treatment naïve, histologically confirmed prostate cancer.

The primary objective of this study is to compare the diagnostic accuracy of T2 weighted imaging (T2WI) and restriction spectrum imaging (RSI) (T2WI + RSI) to that of multiparametric MRI (mpMRI), for the detection of individual prostate cancer foci. Results will be validated against histopathologic findings at prostatectomy as the reference standard.

We hypothesize that T2WI + RSI will detect more clinically significant prostate cancer foci (any Gleason grade group > 2) compared to mpMRI when one-to-one matching between imaging and prostatectomy findings is performed.

Secondary Objectives

-To perform a pilot study evaluating T2WI+RSI/US fusion guided biopsy compared to mpMRI/US fusion biopsy for the diagnosis of clinically significant cancer (any Gleason grade group > 2) in a cohort of patients scheduled for clinically indicated MRI/US fusion guided biopsy. In this pilot study, we hypothesize that RSI/US fusion guided biopsy will be non-inferior to mpMRI/US fusion guided biopsy in the detection of clinically significant prostate cancer.

Primary Objectives:

* To acquire high frequency transrectal microultrasound data in patients undergoing clinically indicated MRI/US fusion guided biopsy.
* To perform additional comparative analyses of mpMRI and RSI images, including analyzing variations in tumor contours between imaging data sets.

ELIGIBILITY:
-Inclusion Criteria:

Primary Objective Cohort

* Treatment naïve patients with histologically confirmed clinically significant prostate cancer (defined as Gleason score > 3+4 and a maximum cancer core length of > 4mm (42)) with a clinical indication for prostate mpMRI for pre-treatment tumor detection and staging
* Patients with anticipated clinical follow-up who are anticipated to undergo surgery at MD Anderson.

Secondary Objective Cohort

* Treatment naïve patients with histologically confirmed intermediate risk prostate cancer (defined as Gleason score > 3+4 and a maximum cancer core length of > 4mm (42)) with a clinical indication for prostate mpMRI, who are to undergo target selection for fusion guided biopsy.
* Patients who are anticipated to undergo fusion guided biopsy at MD Anderson.

Exclusion Criteria:

* Patients who have already received androgen deprivation therapy or undergone prior surgery, radiotherapy or focal ablative therapies to the prostate
* Patients whose weight exceeds 400 pounds
* Patients allergic to gadolinium
* Patients with pacemakers or other implantable devices or conditions that are a contraindication to MRI
* Patients with conditions precluding MR imaging at 3T
* Patients less than 18 years of age
* Patients unable to provide informed consent
* Patients unable to tolerate an endorectal coil
* Patients who have undergone prostate biopsy less than 6 weeks prior to their MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the diagnostic accuracy of T2 weighted imaging (T2WI) and restriction spectrum imaging (RSI) (T2WI + RSI) to that of multiparametric MRI (mpMRI), for the detection of individual prostate cancer foci. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aradhana Venkatesan, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org